CLINICAL TRIAL: NCT03691805
Title: Transcranial Direct Current Stimulation as an Intervention in Tobacco Use Disorder: Effects on Consumption and Craving
Brief Title: Transcranial Direct Current Stimulation - Tobacco Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS-TUD
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Tobacco Use Disorder
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Half of the participants will receive transcranial direct current stimulation, while the others will receive sham stimulation.
Who Masked: Participant
Masking Description: Participants will be blinded as to their assigned study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS over rDLPFC (Active Comparator): Participants will receive anodal tDCS (transcranial direct current stimulation) of the right dorsolateral prefrontal Cortex (DLPFC).
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): Participants will receive sham tDCS (transcranial direct current stimulation) of the DLPFC.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: tDCS — The participants will receive anodal tDCS (transcranial direct current stimulation) of the right dorsolateral prefrontal cortex for 20 minutes on five consecutive days.
  Other Names: sooma medical; transcranial direct current stimulation
  Arms: anodal tDCS over rDLPFC
Device: Sham tDCS — The participants will receive sham tDCS (transcranial direct current stimulation) of the dorsolateral prefrontal cortex for 20 minutes on five consecutive days.
  Arms: sham tDCS

SUMMARY:
This study aims to detect how transcranial direct current stimulation (tDCS) affects smokers' inhibitory control, craving and consumption of tobacco goods.

DETAILED DESCRIPTION:
Participating smokers are to receive anodal transcranial direct current stimulation of the right dorsolateral prefrontal cortex (rDLPFC) for 20 minutes on five consecutive days. Neuropsychological tests on inhibitory control and interviews on smoking habits and craving will be applied before and after the first stimulation as well as after the fifth stimulation.

After a follow-up period of three days, smoking behaviour will be assessed in a telephone interview.

Changes in inhibitory control and smoking behaviour will be compared between an active and a sham stimulation group.This way the effects of transcranial direct current stimulation on tobacco use disorder are to be clarified.

ELIGIBILITY:
Inclusion Criteria:

* tobacco use disorder
* normal or correctable eyesight
* sufficient ability to communicate with the investigators, to answer questions in oral and written form
* fully informed consent
* written informed consent

Exclusion Criteria:

* withdrawal of the declaration of consent
* exclusion criteria for tDCS (metal implants in the head, acute eczema, known epilepsy)
* severe internal, neurological or psychiatric comorbidity
* pharmacotherapy with psychoactive substances within the last 14 days
* axis-I disorder according to ICD-10 and DSM 5 (except tobacco use disorder)
* positive urin drug screening (cannabis, amphetamine, opiates, benzodiazepines, cocaine)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Reduced number of cigarettes smoked | First assessment on Day 1, second on Day 8
  Smoking habits will be assessed via interview at the beginning of the study and after a follow-up period of three days. Number of cigarettes smoked will be compared longitudinally and between groups.

SECONDARY OUTCOMES:
Reduced Carving | First assessment on Day 1, second on Day 5, third on Day 8
  Craving will be assessed using visual analog scales on the first and fifth day of the study as well as in the follow-up interview. Ratings will be compared longitudinally and between groups..
Increased inhibitory control | First and second testing on Day 1, third testing on Day 5
  Inhibitory control will be assessed in neuropsychological tests (Go / No-Go, Stop-Signal Task) before and after the first stimulation session and after the fifth session. Results will be compared longitudinally and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Principal Investigator — ZI Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany

REFERENCES:
- [Derived] Muller T, Shevchenko Y, Gerhardt S, Kiefer F, Vollstadt-Klein S. The influence of perceived stress and self-control on efficacy of repeated transcranial direct current stimulation in non-treatment-seeking smokers. Drug Alcohol Depend. 2021 Sep 1;226:108861. doi: 10.1016/j.drugalcdep.2021.108861. Epub 2021 Jun 24. PMID 34198135